CLINICAL TRIAL: NCT07354555
Title: Discovery And Validation Of New Biomarkers In The Context Of Multiple Myeloma Extramedulary Disease
Brief Title: Multiple Myeloma Extramedulary Disease Samples FFPE
Acronym: MMExFFPE
Status: Not yet recruiting | Type: Observational
Sponsor: BIWAKO (Industry)
Responsible Party: Sponsor
Other Study IDs: BWK-P035
Record Dates: First submitted 2025-11-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma Survival Outcome; Multiple Myeloma and Malignant Plasma Cell Neoplasms
Keywords: Myeloma; Extramedullary disease; histopathology; biomarker
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The study plans to collect formalin fixed embedded samples (FFPE) and to cut unstained histopathological slides for immpunohistochemistry techniques. No DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FFPE Blocks: Samples obtained from patients with multiple myeloma extramedullary disease. The samples should be obtained in the extramedullary disease.

SUMMARY:
This observational study aims to evaluate the feasibility of assembling a retrospective cohort of formalin-fixed paraffin-embedded (FFPE) tissue samples from patients with extramedullary multiple myeloma, together with their associated clinical and pathological data. The study will determine whether these archived samples are suitable for exploratory biomarker assessment.

No intervention is performed. All FFPE samples and clinical data originate exclusively from routine diagnostic procedures and will be analyzed retrospectively for research purposes.

DETAILED DESCRIPTION:
This retrospective observational study aims to determine the feasibility of assembling a cohort of formalin-fixed paraffin-embedded (FFPE) tissue samples from patients with extramedullary multiple myeloma and linking these materials with associated clinical and pathological data. All samples originate from routine diagnostic procedures performed as part of standard clinical care; no prospective interventions or additional tissue collection are involved.

The study evaluates whether archived FFPE specimens and corresponding clinical information can be systematically identified, retrieved, and abstracted using a predefined standardized workflow. Histopathological review and immunohistochemical markers routinely assessed during diagnostic work-up (CD138, CD56, MUM1, light chains) will be used to confirm the diagnosis and describe tumor features. Feasibility will be defined by the proportion of screened cases for which both adequate FFPE material and sufficient clinical data are available to allow inclusion.

The purpose of the study is to generate a structured dataset enabling future biomarker research and to assess whether the operational workflow used for case identification, data abstraction, and sample processing can be reliably scaled for larger retrospective cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically confirmed extramedullary myeloma (excluding plasmacytoma).
* Availability of a representative FFPE block from a surgical specimen.
* Diagnosis established within the past 10 years.
* Availability of associated clinical and follow-up data.

Exclusion Criteria:

* Patients with plasmacytoma only.
* Insufficient or non-representative FFPE material.
* Missing key diagnostic or clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with extramedullary myeloma (excluding plasmacytoma) for whom a representative FFPE block from a surgical specimen was obtained as part of routine clinical care within the past 10 years. Only cases with sufficient clinical, pathological, and follow-up data are included. All samples were collected outside the context of research activities.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of cohort inclusion based on availability of FFPE tissue and confirmed extramedullary disease. | Baseline
  Number of participants who meet both criteria:
  * confirmation of extramedullary disease using predefined clinical and histopathological criteria, and
  * availability of an adequate FFPE tissue block suitable for inclusion.
  Feasibility will be quantified by reporting the proportion of eligible participants among all patients screened for potential inclusion.

SECONDARY OUTCOMES:
Evaluate FFPE analytical quality through expression rates of predefined IHC markers (CD138, CD56, MUM1, light chains). | Baseline
  Percentage of cases showing immunoreactivity for selected markers based on standard immunohistochemistry performed during diagnostic work-up. Marker expression is recorded as positive or negative according to predefined laboratory thresholds.

OTHER OUTCOMES:
Describe the distribution of anatomical sites of extramedullary disease with clinicopathological characteristics of included cases. | Baseline
  Categorization of EMD cases according to the anatomical origin of the archived tissue sample (e.g., soft tissue, liver, CNS, lymph node). Measurement is performed by reviewing sample metadata recorded at the time of diagnostic tissue processing.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Rashed, Principal Investigator — MEDARKRO
Locations (1):
- BIWAKO, Lyon 06, France

IPD SHARING:
Plan to Share IPD: No